CLINICAL TRIAL: NCT01910701
Title: Extension Study of the Family Spirit Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ADHS12-014900
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Parenting
Keywords: Home visiting interventions; American Indian; Community based participatory research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family Spirit Intervention (Experimental): The Family Spirit intervention consists of 52 sessions (30-60 minutes in duration) delivered during a 39-month intervention phase and designed to positively impact a number of maternal and child behavioral and health outcomes.
  Interventions: Behavioral: Family Spirit

INTERVENTIONS:
Behavioral: Family Spirit — The Family Spirit intervention consists of 52 sessions (30-60 minutes in duration) delivered during a 39-month intervention phase and designed to positively impact a number of maternal and child behavioral and health outcomes.

SUMMARY:
The aim of the proposed research is to implement and evaluate a follow-up study of the impact of the Family Spirit family strengthening program among a high-risk sample of Apache mothers and their children. The Family Spirit intervention is a 52-session home-visiting curriculum administered by American Indian paraprofessionals to young mothers from 28 weeks gestation through the child's first 3 years of life. In a series of pilot studies and a recently completed randomized controlled trial, the Family Spirit intervention has been found to positively impact several maternal, parenting and child outcomes up through three years postpartum. In the proposed study, the investigators will implement the Family Spirit intervention to young mothers (12-20 years at conception), with revisions to several assessment measures and to the curriculum such that the substance abuse prevention curriculum modules will be taught earlier than in the original study.

DETAILED DESCRIPTION:
This is a single group pre-post study designed to evaluate the impact of a home visiting intervention in improving parenting self-efficacy and a number of other maternal and child health and behavioral outcomes among a sample of young mothers, including maternal substance use. The Family Spirit intervention consists of 52 sessions (30-60 minutes in duration) delivered during a 39-month intervention phase. All sessions are designed to be taught at the participant's home, but they may also occur at another location chosen by the participant (e.g. study office, vehicle). Outcome data will be collected at Baseline and at 2 months, 6 months, 12 months, 24 months and 36 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant American Indian female less than or equal to 32 weeks gestation.
* Reside within 60 miles of Whiteriver Indian Health Service unit.
* Age 12-20 years of age at time of conception

Exclusion Criteria:

* Completed previous randomized controlled trial of Family Spirit
* ≤11 years old or ≥21 years old at time of conception of index pregnancy.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2013-01; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Increase in score on parenting self-efficacy scale | 24 months postpartum

SECONDARY OUTCOMES:
Improved prenatal and infant medical care practices | 24 months postpartum
  Includes: prenatal care utilization, prenatal use of alcohol/drugs, preconception care, inter-birth intervals, screening for maternal depressive symptoms, breastfeeding, well-child visit utilization, maternal and child health insurance status
Reduction in emergency department visits due to childhood injuries | 24 months postpartum
  Includes: visits for children to emergency department for all causes and due to injury, home safety
Improved school readiness scores | 24 months postpartum
  Includes: parent support for children's learning and development, parent knowledge of child development, parenting behaviors, parent-child relationship, parent stress, child's communication and literacy, child's cognitive skills, child's approach to learning, child's social behavior, and child's physical health and development
Improved score on family economic self-sufficiency scale | 24 months postpartum
Increased referrals for community resources | 24 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, MPH, MA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No